CLINICAL TRIAL: NCT07185620
Title: Effects of Impacted Mandibular Third Molar Surgery Performed With Piezoelectric and Conventional Rotary Systems on Postoperative Sequelae and Quality of Life
Brief Title: Piezoelectric and Conventional Rotary Techniques in Third Molar Surgery: Postoperative Outcomes and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izzet Acikan (Other)
Responsible Party: Sponsor-Investigator, Izzet Acikan, Assistant Professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HRÜ/25.07.46
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Third Molar Extraction; Piezoelectric Technique
Keywords: Third molar; Piezoelectric; Conventional Rotary Systems; Postoperative Sequelae; OHIP-14

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezoelectric Surgery group (Experimental): The group in which osteotomy during third molar extraction was performed using a piezoelectric device.
  Interventions: Procedure: Third molar surgery with piezoelectric system
- Conventional Rotary Systems (Active Comparator): The group in which osteotomy during third molar extraction was performed using a conventional rotary system.
  Interventions: Procedure: Third molar surgery with Conventional Rotary System

INTERVENTIONS:
Procedure: Third molar surgery with piezoelectric system — For the surgical removal of the third molar with a mucoperiosteal flap, osteotomy was performed using a piezoelectric system under continuous irrigation. The mucoperiosteal flap was then repositioned and closed primarily with sutures.
  Arms: Piezoelectric Surgery group
Procedure: Third molar surgery with Conventional Rotary System — For the surgical removal of the third molar with a mucoperiosteal flap, osteotomy was performed using a conventional rotary system under continuous irrigation. The mucoperiosteal flap was then repositioned and closed primarily with sutures.
  Arms: Conventional Rotary Systems

SUMMARY:
This study is a prospective, randomized clinical trial comparing recovery after the surgical removal of impacted lower wisdom teeth. The aim is to evaluate swelling, pain, mouth opening, and quality of life after surgery.

The study was approved by the Ethics Committee of Harran University, and all patients gave written informed consent. It was conducted at the Faculty of Dentistry, Kahramanmaraş Sütçü İmam University. A total of 50 patients participated. They were randomly assigned to two groups: one treated with a piezoelectric device (study group) and the other with a conventional rotary handpiece (control group). All surgeries were performed by the same surgeon under local anesthesia.

In both groups, the tooth was removed, the bone edges were smoothed, the area was cleaned with sterile solution, and the gum flap was closed with stitches. In the piezoelectric group, the bone was removed using an ultrasonic piezoelectric system. In the conventional group, bone removal was performed with a surgical drill under irrigation.

After surgery, patients were followed for pain, swelling, mouth opening, and quality of life. Pain was measured daily for 7 days using a 10-point visual scale (0 = no pain, 10 = worst pain). Mouth opening was measured before surgery, on the 2nd day, and on the 7th day after surgery. Swelling was measured using 3-dimensional facial scans taken before surgery, and on the 2nd and 7th days after surgery. Quality of life was assessed with a short questionnaire (OHIP-14), completed before surgery and on days 2, and 7 after surgery. Higher scores meant a worse impact on daily life.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being over 18 years of age,
* having an indication for impacted third molar extraction in the mandible,
* absence of acute pericoronitis or any other active infection,
* willingness to participate in the study.

Exclusion Criteria:

* Individuals with systemic conditions such as
* diabetes mellitus,
* immunodeficiency,
* bleeding disorders,
* dyspepsia or
* those classified as heavy smokers (over 10 cigarettes daily)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
mouth opening measurement | Maximum mouth opening measurements were performed at three different time points: before surgery, on the 2nd postoperative day, and on the 7th postoperative day, and were recorded in millimeters.
Pain Assessment | Preoperative 20 minutes before local anesthesia administration, postoperative day 1, day 2, day 3, day 4, day 5, day 6, and day 7.
  The patients' pain levels were evaluated using a 10-unit Visual Analog Scale (VAS). The patients were given a form on which they could mark the pain they felt as a score between 0 (no pain) and 10 (the most severe pain) at the following time points: 20 minutes before local anesthesia administration, and on postoperative day 1, day 2, day 3, day 4, day 5, day 6, and day 7. After completing these forms, the patients returned them at the end of the 7th day.
swelling measurement | For the measurement of swelling, each patient underwent three-dimensional facial scanning at three time points: immediately before surgery (T0), on the 2nd postoperative day (T1), and on the 7th postoperative day (T2).
  To objectively evaluate postoperative facial swelling, a 3D facial scanning method was employed. All facial scans were performed in the same room, with a standardized position and similar lighting conditions. To obtain three-dimensional facial images, the Qlone application (EyeCue Vision Technologies LTD.) running on an iPhone 14 device equipped with TrueDepth technology was used. This smartphone-based application provides a guided scanning procedure that enables a rapid and detailed capture of the patient's face. At the end of each scanning session, an STL file representing the patient's facial structure was generated. The obtained STL-format facial models were imported into the 3D imaging software 3D Slicer. T0 and T1/T2 facial scans were superimposed within 3D Slicer to detect changes occurring in the facial surface. The superimposition process was carried out using surface registration, referencing stable anatomical regions of the face.
Quality of Life Assessment | Oral health-related quality of life was evaluated using the OHIP-14. Participants completed the questionnaire preoperatively, and on postoperative days 2 and 7.
  Quality of life was evaluated before and after surgery using the OHIP-14 questionnaire. The OHIP-14 assessment was performed preoperatively, and on postoperative days 2 and 7. Each question was rated on a 4-point scale: 1 = "never," 2 = "sometimes," 3 = "fairly often," and 4 = "very often." The possible total score ranged from 0 to 56, with higher scores reflecting greater impairment in quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Faculty of Dentistry, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cantore S, Silva FFVE, Bizzoca ME, Smimmo A, Lo Muzio L, Vianna Camolesi GC, Perez-Sayans M, Ballini A. Enhancing Lower Third Molar Surgery: Using The Piezoelectric Technique for Superior Postoperative Outcomes and Complication Prevention. Dent J (Basel). 2024 Nov 1;12(11):353. doi: 10.3390/dj12110353. PMID 39590403
- [Background] Erdem MK, Cambazoglu M. A comparative analysis of postoperative morbidity and alveolar bone regeneration following surgical extraction of impacted lower third molar teeth using piezosurgery and conventional instruments: a split-mouth clinical investigation. Eur J Med Res. 2024 Sep 14;29(1):460. doi: 10.1186/s40001-024-02051-8. PMID 39272144
- [Background] Demirci A, Bayram F, Dergin G. Piezosurgery versus conventional rotary surgery for impacted third molars: A randomised, split-mouth, clinical pilot trial. Med Oral Patol Oral Cir Bucal. 2024 Jan 1;29(1):e1-e8. doi: 10.4317/medoral.25929. PMID 37992138